CLINICAL TRIAL: NCT05930977
Title: Outcomes of Thyroid Auto Transplantation Following Total Thyroidectomy in Benign Thyroid Disorders Protocol
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohamed Aly Hamam, Mahmoud Mahamed Aly, Sohag University
Other Study IDs: Soh-Med-23-06-04MS
Record Dates: First submitted 2023-06-15; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Thyroid Diseases
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient undergone total thyroidectomy followed by thyroid auto transplantation
  Interventions: Procedure: total thyroidectomy followed by thyroid auto transplantation

INTERVENTIONS:
Procedure: total thyroidectomy followed by thyroid auto transplantation — All studied cases received general endotracheal anaesthesia, and all underwent total thyroidectomy.
  Frozen section will be done intraoperative to exclude malignancy and obtain piece of healthy tissue part .
  Most healthy-looking part of gland was selected after complete excision. Thyroid tissue to be transplanted weighed between two and five grammes. This section was finely split into ten-fifteen fragments with scalpel. Small pocket was created in sternomastoid muscle, into which these minor fragments were implanted, and this pocket was closed with absorbable sutures to prevent displacement of implanted fragments and was marked with metallic stables, as well as good hemostasis of thyroid bed and skin was closed with subcuticular sutures using absorbable three-zero Vicryl sutures.

SUMMARY:
the study aimed at evaluating efficacy of auto-transplantation of thyroid tissue after total thyroidectomy in benign thyroid disorders to keep the patient euthyroid with no need for life long hormone replacement therapy.

DETAILED DESCRIPTION:
This study will be a prospective study which will be conducted at Sohag University Hospital after approval of the protocol the study population include . Adult patients with goiters are seen in the general surgery outpatient clinic The study included thirty studied cases presented in the outpatient clinic with benign thyroid disorders for whom total thyroidectomy was performed

ELIGIBILITY:
Inclusion Criteria:

* Patients proved to have benign thyroid disorders operable and candidate for total thyroidectomy Adult patients who agreed and consented to do the procedure.

Exclusion Criteria:

* Patients with high suspicion of malignancy , unfit and refused the procedure

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with benign multi nodular goiter
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Thyroid function following thyroid auto transplantation after total thyroidectomy | six months
  Thyroid hormone levels will be assessed after auto transplantation of thyroid tissue from benign thyroid patients following total thyroidectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No